CLINICAL TRIAL: NCT02705521
Title: A Multi-centre, Randomised, Controlled Study Comparing Gamification With Remote Monitoring Against Standard Rehabilitation, for Patients After Arthroscopic Subacromial Decompression Surgery
Brief Title: Comparing Gamification With Remote Monitoring Against Standard Rehabilitation, for Patients After Arthroscopic Subacromial Decompression Surgery
Acronym: GAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Northern Care Alliance NHS Foundation Trust (Other); Royal Bolton Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 179371
Record Dates: First submitted 2016-03-05; First posted 2016-03-10 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Shoulder Impingement Syndrome; Subacromial Impingement Syndrome
Keywords: shoulder; impingement; rehabilitation; physiotherapy; gamification; activation; engagement
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as usual group (No Intervention): Patients will attend physiotherapy on a weekly basis for assessment (standard physiotherapy). They will be assessed for progression and be provided with a home exercise program. Range of motion in their shoulder will be collected on a weekly basis using the MIRA technology. Patients will be required to complete an exercise diary documenting the exercises performed as well as duration and frequency.
- Treatment as usual plus Exergames group (Experimental): Patients will attend physiotherapy on a weekly basis for assessment (standard physiotherapy). Rather than use a home exercise program patients will be provided with a laptop computer and kinect sensor. they will use the new technology to play 'Exergames' each program will be tailored to the patients progress and patients can play the system as often as they wish. Patients will be required to complete an exercise diary documenting the exercises performed as well as duration and frequency.
  Interventions: Device: Exergames- Laptop and MIcrosoft Kinect

INTERVENTIONS:
Device: Exergames- Laptop and MIcrosoft Kinect — Following surgery each patient will have a set of games for them to play using their affecting shoulder. These games have been designed by physiotherapists and shoulder surgeons to improve the functional range of movement in their shoulder
  Other Names: Microsoft Kinect; MIRA Rehab
  Arms: Treatment as usual plus Exergames group

SUMMARY:
This randomised prospective controlled trial will investigate patients with impingement syndrome who undergo arthroscopic subacromial decompression. The intervention group will receive physiotherapy aided by automated sensor-based technology which will help them perform exergames and track their rehabilitation progress. The control group will be treated by standard physiotherapy protocols. The two groups will be compared using patient reported outcome measures and assessment of shoulder range of movement before and after the shoulder surgery.

Data will be collected on patient experience, engagement with the rehabilitation process and the usability of the sensor-based technology through the use exergames. This will guide development of methods to quantify patient activation and engagement.

Hypothesis:

1. There will be a significant clinical difference in post-surgical improvement measured by patient reported outcomes when physiotherapy is aided by automated sensor-based technology to perform Exergames and track progress, compared to standard physiotherapy protocols.
2. There will be a significant difference in post-surgical improvement in range of shoulder movement and patient improvement, measured by patient reported out-comes when physiotherapy is aided by automated sensor-based technology to perform exergames and track progress, compared to standard physiotherapy protocols.

DETAILED DESCRIPTION:
Background:

Musculoskeletal problems are one of the most common reasons for seeking medical advice, with estimates of up to 20% of adults annually consulting their general practitioner. The prevalence of shoulder problems in the population is approximately 2.5%(Jordon et al 2010). In 2012/13, there were over 7.1 million outpatient appointments for trauma and orthopaedics in England (accounting for 9.3% of all outpatient attendances) and over 4 million of these visits were followup after the initial consultation (Hospital Episode Statistics). The average cost for each outpatient follow up is £76. At a time when the NHS is under considerable financial burden we are constantly looking at ways and means of reducing the number of outpatient appointments and the length of time for which a patient required followup. By improving rehabilitation protocols patients may complete their recovery more rapidly which may reduce clinician patient face-to-face interactions. This may free up this valuable resource which can be directed towards more complex clinical requirements.

Patient Engagement:

One of the major factors that influence patient outcomes is their engagement with the rehabilitation program.

Rehabilitation professionals have long suspected that a patient's motivation plays an important role in determining the outcome of therapy, despite the lack of a clear definition of the phenomenon (Maclean et al. 2002). It is estimated that up to 65% of patients are non/partially adherent to their home exercise program (Meichenbaum 1987). Classically, patients have completed home exercise diaries. However, studies have suggested that these are often completed retrospectively. This may encourage patients to exaggerate the amount of activity performed. Hoelscher at al (1984), timed patients at home performing a relaxation exercise program and compared this to patient reported duration. They found that the latter tended to suggest a higher level of adherence. The Exergames programmes actively track patient interaction with the software. Each activity records the length of interaction, progress through rehabilitation allowing the clinician to have a clearer indication of patient engagement in rehabilitation.

Patient activation describes the knowledge, skills and confidence a person has in managing their own health and health care. Intervening to increase activation can improve a patient's engagement and health outcomes. This is an important factor in helping patients manage their health (Kings Fund 2015). As a part of this study we will quantify patient engagement. Through this we can develop and validate a new tool to comprehensively measure patient outcomes using four domains. These will be Patient reported pain and function (P), shoulder range of movement i.e.

Kinematics (K), patient activation or engagement (E) and patient experience (X).

Gamification:

Traditional evaluation of the patient's range of motion usually occurs in a clinic, often using subjective and informal methods of angle measurement. This has the potential to create discrepancies in findings between clinicians. To reduce the use of healthcare resources, make the clinical assessment more convenient for the patient, to improve the quality of the information collected and the assessment conducted, electronic measurement has the potential to perform repeatable validated objective results.

If combined with appropriate principles of gamification, these measurements can become a part of the rehabilitation process with potentially faster clinical improvement and comprehensive analysis of patient generated outcomes. In light of this, there has been a wave of support for the implementation of gaming elements in healthcare technologies.

'Gamification' involves the incorporation of game mechanics in a non-game setting and a tailored user interface for better learning which encourages engagement (King 2013). Reward systems, competition and immediate feedback improve user experience and have been implemented in healthcare related fields where patients have become a niche target group (Lin 2013). This may in turn increase patient activation allowing them to manage their own health.

MIRA:

MIRA Rehab is a company who has developed software designed for the rehabilitation of medical conditions.

Combined with a Microsoft Kinect sensor it accurately traces the range of motion in the shoulder. MIRA uses games which are built based upon the best clinical practice and expertise from specialist clinicians. The MIRA programme enables patients to progress through different levels within the games whilst engaging in their rehabilitation programme.

Research Design and Methodology:

Methodology:

90 patients will be recruited to a 3 month rehabilitation programme following a standard subacromial decompression

+/biceps tenotomy for impingement syndrome. Patients will be randomised into two groups:

1. Standard postoperative physiotherapy regime without the use of accessory software (Treatment as usual Group).
2. Postoperative regime of physiotherapy plus Exergames utilizing principles of gamification.

Power calculation:

A sample size calculation was performed using Oxford Shoulder Score (OSS) sample data collected on patients previously undergoing arthroscopic subacromial decompression. [Alpha error set at 0.05, and beta error at 0.8, mean difference of 5 points12 in the OSS, standard deviation 6.96] Based upon this, a sample size of 32 patients in each group would be required.

A second sample size calculation was performed based on the disabilities of arm shoulder and hand (DASH) outcome measure. [Alpha error set at 0.05, and beta error at 0.8, mean difference of 15 points in the DASH13, standard deviation 23] Based upon this, a sample size of 37 patients in each group would be required.

Therefore, a target of 45 patients per group was chosen to allow for some participants withdrawing from the study (20%).

Treatment as usual Group:

Patients will attend physiotherapy on a weekly basis for assessment. They will be assessed for progression and be provided with a home exercise program. Range of motion in their shoulder will be collected on a weekly basis using the MIRA technology. Patients will be required to complete an exercise diary documenting the exercises performed as well as duration and frequency.

Treatment as usual plus Exergames Group:

Prior to commencing the study the physiotherapists will set up and initially demonstrate the Exergames to the intervention participants in the home setting. This will ensure the safety of the patients and address any technological issues that may arise. Patients will attend physiotherapy on a weekly basis as well as partaking in a set of tailored Exergames to play in the home system. The MIRA software will record the patient engagement with the system including number of sessions and duration of play. Patients will also be asked to complete an exercise diary.

VISIT SUMMARY

Baseline (Clinic Consultation):

Patient's eligibility to participate in the study will be assessed; inclusion/ exclusion criteria must be met. The Patient Information Sheet will be given to the patient when they are listed for surgery. Prior to their surgery date, the patient will be contacted by a member of the research team, to see if they would like to participate in the study. Patient will be asked to give their consent to the study on the day of surgery. Past medical history will be reviewed and patient demographics will be documented. Relevant questions and scoring will be taken for baseline reference.

+ 24 hours (following baseline assessments) The patient reported outcome measures questionnaires will be repeated by all patients.

Day 1 Patient attends hospital for surgical treatment. Confirmation of study consent must be confirmed. A study diary will be dispensed to patient. Study coordinator will give full explanation regarding completion of the diary.

Day 7,14,21,28,35,42,49,56,63,70,77.

Patient must attend physiotherapy clinic at day 7,14,21,28,35,42,49,56,63,70,77. A scheduled visit window to allow flexibility is +/- 2 days. Patient is to continue with their post-operative physiotherapy regime depending on the treatment group they have been randomised. Range of Movement will be assessed and documented by the research physiotherapist. Each patient diary will be reviewed and assessed.

Day 84/85 Patient diary will be reviewed and returned. On completion of the 12 week programme all patients (N=90) will complete all outcome questionnaires, Patients randomised to Exergames arm will complete a Systems Usability score for the MIRA software. Range of movement will be recorded by MIRA and documented by the research physio-therapist.

Day 365 One year post surgery all patients (N=90) will complete the scoring questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of impingement syndrome based upon history, clinical examination and radiological findings that require arthroscopic subacromial decompression.
2. The patient has access to the internet to allow for the remote monitoring element of the intervention.
3. The patient needs to be able to use the sensor based technology safely, as judged by the research team.
4. The patient is willing to consent to follow-up over a twelve month period.
5. The patient has capacity to consent to the study.

Exclusion Criteria:

1. Aged less than 18 or greater than 70
2. Patients who are unwilling or unable to consent
3. Previous arthroscopic shoulder surgery
4. Patients undergoing radiotherapy
5. Patients with type 1 or type 2 diabetes
6. Patients not fit for general anaesthetic
7. Patients with significant cardiac dysfunction
8. Uncontrolled hypertension
9. Acute illness
10. History of stroke / neuromuscular conditions preventing the use of Exergames
11. Patient is currently enrolled in another clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Oxford shoulder score | 3 months and twelve months
  Patients will be assessed for a significant difference in the OSS at 3 at 12 months compared with the treatment as usual group.

SECONDARY OUTCOMES:
The Disabilities of the Arm, Shoulder and Hand score | 3 months and 12 months
  Patients will be assessed for a significant difference in the DASH score at 3 at 12 months compared with the treatment as usual group.
The European Quality of Life 5 Dimensions (EQ5D) | 3 months and 12 months
  Patients will be assessed for a significant difference in the EQ5D at 3 at 12 months compared with the treatment as usual group.
Visual analogue Scale for pain (VAS) | 3 months and 12 months
  Patients will be assessed for a significant difference in the EQ5D at 3 at 12 months compared with the treatment as usual group.
Shoulder range of movement | 3 months
  Patients will be assessed using the MIRA software to see if there is a statistically significant difference in the cardinal ranges of motion in the shoulder joint

CONTACTS AND LOCATIONS:
Overall Officials: Bibhas Roy, MB CHB MSC, Principal Investigator — Central Manchester University Hospitals Trust
Locations (3):
- United Kingdom (3):
  - Royal Bolton Hospital, Bolton, Lancashire
  - Trafford General Hospital, Manchester, Lancashire
  - Salford Royal Hospital, Manchester, Lancashire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bigliani LU, Ticker JB, Flatow EL, Soslowsky LJ, Mow VC. The relationship of acromial architecture to rotator cuff disease. Clin Sports Med. 1991 Oct;10(4):823-38. PMID 1934099
- [Background] Kuhn JE. Exercise in the treatment of rotator cuff impingement: a systematic review and a synthesized evidence-based rehabilitation protocol. J Shoulder Elbow Surg. 2009 Jan-Feb;18(1):138-60. doi: 10.1016/j.jse.2008.06.004. Epub 2008 Oct 2. PMID 18835532
- [Background] Jordan KP, Kadam UT, Hayward R, Porcheret M, Young C, Croft P. Annual consultation prevalence of regional musculoskeletal problems in primary care: an observational study. BMC Musculoskelet Disord. 2010 Jul 2;11:144. doi: 10.1186/1471-2474-11-144. PMID 20598124
- [Background] Olley LM, Carr AJ. The use of a patient-based questionnaire (the Oxford Shoulder Score) to assess outcome after rotator cuff repair. Ann R Coll Surg Engl. 2008 May;90(4):326-31. doi: 10.1308/003588408X285964. PMID 18492399
- [Background] Maclean N, Pound P, Wolfe C, Rudd A. The concept of patient motivation: a qualitative analysis of stroke professionals' attitudes. Stroke. 2002 Feb;33(2):444-8. doi: 10.1161/hs0202.102367. PMID 11823650
- [Background] King D, Greaves F, Exeter C, Darzi A. 'Gamification': influencing health behaviours with games. J R Soc Med. 2013 Mar;106(3):76-8. doi: 10.1177/0141076813480996. No abstract available. PMID 23481424
- [Background] Lin RJ, Zhu X. Leveraging social media for preventive care-A gamification system and insights. Stud Health Technol Inform. 2012;180:838-42. PMID 22874310
- [Background] Cloke DJ, Watson H, Purdy S, Steen IN, Williams JR. A pilot randomized, controlled trial of treatment for painful arc of the shoulder. J Shoulder Elbow Surg. 2008 Jan-Feb;17(1 Suppl):17S-21S. doi: 10.1016/j.jse.2007.07.005. PMID 18069016
- [Background] Dawson J, Fitzpatrick R, Carr A. Questionnaire on the perceptions of patients about shoulder surgery. J Bone Joint Surg Br. 1996 Jul;78(4):593-600. PMID 8682827
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172